CLINICAL TRIAL: NCT04401085
Title: Herd Immunity Study SARS-CoV-2-CZ-Preval
Brief Title: COVID-19: Herd Immunity Study in the Czech Republic
Acronym: SARSCoV2CZPrev
Status: Completed | Type: Observational
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: Ministry of Health, Czech Republic (Other Government); Palacky University (Other); Masaryk University (Other); University of Ostrava (Other); Faculty of Military Health Sciences, University of Defence in Brno (Unknown); Faculty of Health Studies, J. E. Purkyně University in Ústí nad Labem (Unknown); Charles University, Czech Republic (Other); Institute for Clinical and Experimental Medicine (Other Government); General University Hospital, Prague (Other); University Hospital Olomouc (Other); Brno University Hospital (Other); Krajská zdravotní, a.s., Ústí nad Labem Region Hospitals (Unknown); Military University Hospital, Prague (Other); Masaryk Memorial Cancer Institute (Other); Czech Academy of Sciences (Other); Czech Statistical Office (Unknown)
Responsible Party: Sponsor
Other Study IDs: UZIS 2020/1
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: COVID; SARS-CoV 2
Keywords: SARS-CoV-2; prevalence; asymptomatic infection; spread dynamics
MeSH Terms: conditions — Asymptomatic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Only in one region, venous blood sampling will be archived in the biobank for subsequent quantitative analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Population area cohort - Control Cohort: A population cohort of asymptomatic individuals (only adults). This is a representative sample of the population, which are part of the research project of Institute for Clinical and Experimental Medicine and Czech Academy of Sciences. The second subsample included individuals from the official household survey of Czech Statistical Office. This cohort allowed better comparative analysis of other population cohorts from specific geographical areas.
  Interventions: Diagnostic Test: SARS-CoV-2 diagnostic rapid test
- Population cohort from specific geographical areas: This cohort is based on epidemiologically defined demographic parameters. These are populations from the following geographical areas:
  Brno and the South Moravian Region; Praha; Olomouc; Litoměřice; Litovel and Uničov.
  Interventions: Diagnostic Test: SARS-CoV-2 diagnostic rapid test; Diagnostic Test: Quantitative analysis of SARS-CoV-2 antibodies
- Chronically ill patients cohort: A cohort of chronically ill people enrolled by Institute for Clinical and Experimental Medicine with chronic cardiovascular problems, hypertension, or diabetes.
  Interventions: Diagnostic Test: SARS-CoV-2 diagnostic rapid test

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 diagnostic rapid test — The rapid test detects the presence of antibodies against SARS-CoV-2 in the IgM and IgG class by the immunochromatographic reaction. It cannot detect early infection, the antibodies will probably appear two weeks after possible infection. The collection will be performed by finger puncture.
Diagnostic Test: Quantitative analysis of SARS-CoV-2 antibodies — The subsample from Olomouc region (Olomouc, Uničov, Litovel) is based on venous blood sampling and archiving for subsequent quantitative analysis of SARS-CoV-2 antibodies. These tests detect immunoglobulins M and G (IgM and IgG).
  Groups: Population cohort from specific geographical areas

SUMMARY:
The aim of the SARS-CoV-2-CZ-Preval study is to quantify the prevalence of individuals with a history of SARS-CoV-2 coronavirus infection in the Czech population, except for those diagnosed with COVID-19 by methods based on direct detection of SARS-CoV- 2, including individuals with a subclinical course of the disease.

DETAILED DESCRIPTION:
COVID-19 is caused by a new type of coronavirus called SARS-CoV-2. It is a highly infectious disease, manifested mainly by fever, respiratory problems, muscle pain, and fatigue. However, despite the publication of hundreds of papers in the literature, fundamental information about the spread and course of the disease is still lacking in COVID-19. One of such key pieces of information is the prevalence of asymptomatic individuals with SARS-CoV-2 infection, which has a significant effect on the dynamics of the spread of COVID-19 in the Czech Republic and within individual regions and localities.

The SARS-CoV-2-CZ-Preval study is aiming at quantification of the prevalence of individuals with a history of SARS-CoV-2 coronavirus infection in the Czech population, except for those diagnosed with COVID-19 by methods based on direct detection of SARS-CoV- 2, including individuals with a subclinical course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* signed Informed Consent
* residing in The Czech Republic
* demographic criteria: (i) persons aged 8-17 (specific children's cohort), (ii) persons aged 18-89
* clinical criteria: (i) without acute health problems (ii) without a confirmed diagnosis of COVID-19
* geographic criteria: according to a particular cohort definition

Ages: 8 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population area cohort is chosen based on random selection. The cohort from specific demographic areas are volunteers from the regions described in the cohort. The population of chronically ill people is a cohort enrolled by Institute for Clinical and Experimental Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 27000 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Estimation of the actual prevalence of SARS-CoV-2 positive persons in the Czech Republic. | May 2020
  Statistically, the primary objective is formulated as an estimate of the cumulative prevalence of SARS-CoV-2 positive individuals in geographically defined subpopulations of the Czech Republic with declared reliability of +/- 2%. For this primary objective, the required sample size in individual geographical cohorts is calculated. The positivity of SARS-CoV-2 individuals who have not been diagnosed with COVID-19 by a standard route of the detection will be assessed by the presence of specific IgM or IgG antibodies in the blood (antibody tests).

SECONDARY OUTCOMES:
Estimation of the proportion of people with a subclinical course of the disease | May 2020
  The proportion of SARS-CoV-2 positive persons who, according to the questionnaire, will not report any or minimal symptoms in the anamnesis.
Estimation of the cumulative prevalence of the disease and the proportion of people with a subclinical course differences between subcohorts according to demographic, social and clinically relevant stratifications. | May 2020
Estimation of the proportion of persons suitable for the donation of convalescent plasma | May 2020
  The estimation will be calculated according to the prevalence of the disease in the population after excluding contraindications to blood donation (age, health status, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Roman Chlíbek, Prof., Study Director — University of Defence in Brno; Rastislav Maďar, Assoc. Prof., Study Director — University of Ostrava, Faculy of Medicine; Marián Hajdúch, Assoc. Prof., Study Director — Institute of Molecular and Translational Medicine; Ladislav Dušek, Prof., Study Director — Institute of Health Information and Statistics of the Czech Republic; Roman Prymula, Prof., Study Chair — Ministry of Health, Czech Republic; Jarmila Rážová, M.D.; Ph.D., Study Chair — Ministry of Health, Czech Republic; Věra Adámková, Prof., Principal Investigator — Institute for Clinical and Experimental Medicine; Aleksi Šedo, Prof., Principal Investigator — Charles University, First Faculty of Medicine; Vladimír Černý, Prof., Principal Investigator — Charles University, Faculty of Medicine in Hradec Králové; Jaroslav Štěrba, Prof., Principal Investigator — Brno University Hospital; David Feltl, Prof., Principal Investigator — General University Hospital, Prague; Martin Repko, Prof., Principal Investigator — Masaryk University, Faculty of Medicine; Dalibor Valík, Prof., Principal Investigator — Masaryk Memorial Cancer Institute; Zdeněk Havel, Assoc. Prof., Principal Investigator — J. E. Purkyně University in Ústí nad Labem, Faculty of Health Studies
Locations (1):
- Institute of Health Information and Statistics of the Czech Republic, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available